CLINICAL TRIAL: NCT02837341
Title: Camera-based Measurement of Respiratory Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EKNZ 2015-306
Record Dates: First submitted 2015-11-12; First posted 2016-07-19 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Tachypnea
Keywords: medical device
MeSH Terms: conditions — Tachypnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Volunteers (Other): Monitoring of respiratory rates via camera-based System Monitoring of respiratory rate by Philips®Vital Sign Device - Camera-based system (Prototype) and capnography simultaneously.
  Interventions: Device: Philips®Vital Sign Device - Camera-based system (Prototype)

INTERVENTIONS:
Device: Philips®Vital Sign Device - Camera-based system (Prototype) — Respiratory rates monitored via camera-based system and capnography simultaneously The "Philips Vital Sign Device" will record chest movements by camera. The program will use an algorithm to convert the chest movements into the respiratory rate

SUMMARY:
Respiratory rate as an important predictor for adverse events, but still a neglected vital sign.

Precise and simple measurement of the respiratory rate in volunteers by a new electronic camera device in different settings.

DETAILED DESCRIPTION:
Background of the study The respiratory rate (RR) is an important vital sign to be monitored in the emergency room, as it is a sensitive predictor of risk and critical illness . An increased RR is a sensitive and independent marker of increased mortality in patients with community acquired pneumonia and in unselected patients presenting to the emergency department (ED): This is why the RR is a component in many risk scores for prediction of adverse outcomes, such as the 'Confusion/Urea/Respiratory rate/Blood pressure/-Age 65 or older' (CURB-65) score, the Modified Early Warning Score (MEWS), Trauma Score, Revised Trauma Score, APACHE II (Acute Physiology and Chronic Health Evaluation) and PRISM (Paediatric Risk of Mortality ). Additionally, it is part of the Systemic Inflammatory Response Syndrome (SIRS) Sepsis-definition and definitions for weaning a patient from a ventilator (RSBI, Rapid Shallow Breathing Index, ). In some cases, measurement of the oxygen saturation is not sufficient as tachypnoea may not always have a connection to hypoxia . Hence, RR plays an important role in triage of patients presenting to the emergency room. Especially tachypnoea brings the need for more detailed monitoring and investigation. Tachypnea/Bradypnoea can be seen as a red flag and may indicate a big variety of diseases like heart failure, pneumonia, metabolic disturbances or pulmonary embolism. Recent studies could demonstrate that also trends of RR are reliable predictors of clinical outcome. Especially an increase in tachypnoea during hospitalisation is associated with high mortality A careful and exact measurement is essential. In emergency situations the RR is one component of the Emergency Severity Index (ESI) algorithm and a mandatory vital sign measured at decision point "D". However, its measurement is often omitted due to time constraints . Moreover documented pathologic RR in ER scenarios indicating hypoxia are often neglected leading to fatal events and contributing to deaths caused by medical errors.

According to recommendations of the World Health Organization (WHO) the RR should be measured by counting the breaths over a period of 1 minute by counting how many times the chest rises. This should be done when the patient is at rest. This appears impractical due to time consumption and workload for nursing staff in an emergency department. Studies have shown that this fact is a main reason why RR is often not recorded and critical situations might be missed. A prospective study by Lovett et al. demonstrated that the measurement of RR by nursing staff and even by impedance plethysmography as a common used device have a low sensitivity in detecting brady- or tachypnoea. The vital sign measurements may also differ according to observer variability. The approach to use mobile devices for RR measurement has shown encouraging results to improve efficiency in comparison to traditional methods though the field of using mobile devices is still in an experimental stadium.

The investigators aim to compare the results given by the camera-based measurements to the results given by capnography. The goal of the survey is to analyse the accuracy of measurements performed by the software.

The investigators will recruit healthy volunteers without any history of pulmonary diseases for an analysis of RR monitoring. Upon agreement the investigators will measure the RR camera-based by a device and simultaneously count the RR by capnography as a reference method. The data will be collected through a standardised protocol and archived in an Access(R) database. Different settings (e.g. supine vs sitting) will be assessed. Results will be depicted in a Bland-Altmann plot. In a first step the investigators plan to do a feasibility study, after that, as a second step, they will continue to measure the RR in different positions and situations to simulate a situation similar to emergency conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* healthy male volunteers
* BMI 19-25

Exclusion Criteria:

* pulmonary diseases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Absolute difference between respiratory rates at different breathing spectra measured via camera | study day 1
  The study compares respiratory rates obtained by 3 methods. 1. Camera based measurement, 2. with capnography and 3. with the WHO criterion standard of counting breaths for 1 Minute (18 measurements in whole).
  The unit of respiratory rate is breaths per minute (e.g. 18/min) To test the accuracy of the Philips Software investigators will compare the camera-based measurements with the measurements done by capnography (as a gold standard). The statistical results will be depicted in a Bland-Altman-Plot
Absolute difference between respiratory rates at different breathing spectra measured via capnography | study day 1
  The study compares respiratory rates obtained by 3 methods. 1. Camera based measurement, 2. with capnography and 3. with the WHO criterion standard of counting breaths for 1 Minute (18 measurements in whole).
  The unit of respiratory rate is breaths per minute (e.g. 18/min) To test the accuracy of the Philips Software investigators will compare the camera-based measurements with the measurements done by capnography (as a gold standard). The statistical results will be depicted in a Bland-Altman-Plot
Absolute difference between respiratory rates at different breathing spectra measured via WHO standard (counting breaths for one minute) | study day 1
  The study compares respiratory rates obtained by 3 methods. 1. Camera based measurement, 2. with capnography and 3. with the WHO criterion standard of counting breaths for 1 Minute (18 measurements in whole).
  The unit of respiratory rate is breaths per minute (e.g. 18/min) To test the accuracy of the Philips Software investigators will compare the camera-based measurements with the measurements done by capnography (as a gold standard). The statistical results will be depicted in a Bland-Altman-Plot

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nickel, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Intensive Care Unit, University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hodgetts TJ, Kenward G, Vlachonikolis IG, Payne S, Castle N. The identification of risk factors for cardiac arrest and formulation of activation criteria to alert a medical emergency team. Resuscitation. 2002 Aug;54(2):125-31. doi: 10.1016/s0300-9572(02)00100-4. PMID 12161291
- [Result] Strauss R, Ewig S, Richter K, Konig T, Heller G, Bauer TT. The prognostic significance of respiratory rate in patients with pneumonia: a retrospective analysis of data from 705,928 hospitalized patients in Germany from 2010-2012. Dtsch Arztebl Int. 2014 Jul 21;111(29-30):503-8, i-v. doi: 10.3238/arztebl.2014.0503. PMID 25142073
- [Result] Pollack MM, Ruttimann UE, Getson PR. Pediatric risk of mortality (PRISM) score. Crit Care Med. 1988 Nov;16(11):1110-6. doi: 10.1097/00003246-198811000-00006. PMID 3048900
- [Result] Bone RC, Sprung CL, Sibbald WJ. Definitions for sepsis and organ failure. Crit Care Med. 1992 Jun;20(6):724-6. doi: 10.1097/00003246-199206000-00002. No abstract available. PMID 1597021
- [Result] Meade M, Guyatt G, Cook D, Griffith L, Sinuff T, Kergl C, Mancebo J, Esteban A, Epstein S. Predicting success in weaning from mechanical ventilation. Chest. 2001 Dec;120(6 Suppl):400S-24S. doi: 10.1378/chest.120.6_suppl.400s. PMID 11742961
- [Result] Mower WR, Sachs C, Nicklin EL, Safa P, Baraff LJ. A comparison of pulse oximetry and respiratory rate in patient screening. Respir Med. 1996 Nov;90(10):593-9. doi: 10.1016/s0954-6111(96)90017-7. PMID 8959116
- [Result] Subbe CP, Kruger M, Rutherford P, Gemmel L. Validation of a modified Early Warning Score in medical admissions. QJM. 2001 Oct;94(10):521-6. doi: 10.1093/qjmed/94.10.521. PMID 11588210
- [Result] Goldhill DR, White SA, Sumner A. Physiological values and procedures in the 24 h before ICU admission from the ward. Anaesthesia. 1999 Jun;54(6):529-34. doi: 10.1046/j.1365-2044.1999.00837.x. PMID 10403864
- [Result] Kellett J, Murray A, Woodworth S, Huang W. Trends in weighted vital signs and the clinical course of 44,531 acutely ill medical patients while in hospital. Acute Med. 2015;14(1):3-9. PMID 25745643
- [Result] Grossmann FF, Nickel CH, Christ M, Schneider K, Spirig R, Bingisser R. Transporting clinical tools to new settings: cultural adaptation and validation of the Emergency Severity Index in German. Ann Emerg Med. 2011 Mar;57(3):257-64. doi: 10.1016/j.annemergmed.2010.07.021. Epub 2010 Oct 16. PMID 20952097
- [Result] Venkatesh AK, Curley D, Chang Y, Liu SW. Communication of Vital Signs at Emergency Department Handoff: Opportunities for Improvement. Ann Emerg Med. 2015 Aug;66(2):125-30. doi: 10.1016/j.annemergmed.2015.02.025. Epub 2015 Mar 21. PMID 25805116
- [Result] Hogan J. Why don't nurses monitor the respiratory rates of patients? Br J Nurs. 2006 May 11-24;15(9):489-92. doi: 10.12968/bjon.2006.15.9.21087. PMID 16723921
- [Result] Lovett PB, Buchwald JM, Sturmann K, Bijur P. The vexatious vital: neither clinical measurements by nurses nor an electronic monitor provides accurate measurements of respiratory rate in triage. Ann Emerg Med. 2005 Jan;45(1):68-76. doi: 10.1016/j.annemergmed.2004.06.016. PMID 15635313
- [Result] Edmonds ZV, Mower WR, Lovato LM, Lomeli R. The reliability of vital sign measurements. Ann Emerg Med. 2002 Mar;39(3):233-7. doi: 10.1067/mem.2002.122017. PMID 11867974
- [Result] Karlen W, Gan H, Chiu M, Dunsmuir D, Zhou G, Dumont GA, Ansermino JM. Improving the accuracy and efficiency of respiratory rate measurements in children using mobile devices. PLoS One. 2014 Jun 11;9(6):e99266. doi: 10.1371/journal.pone.0099266. eCollection 2014. PMID 24919062
- [Result] Folke M, Cernerud L, Ekstrom M, Hok B. Critical review of non-invasive respiratory monitoring in medical care. Med Biol Eng Comput. 2003 Jul;41(4):377-83. doi: 10.1007/BF02348078. PMID 12892358